CLINICAL TRIAL: NCT06885372
Title: Long-term Follow up of the Stability 1 Trial
Acronym: STABILITY LTF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 104524
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: LET; ACL Reconstruction; Osteoarthritis (OA) of the Knee
Keywords: ACL; ACL injuries; ACL reconstruction; LET; Osteoarthritis; Knee osteoarthritis; Orthopaedics; Anterolateral ligament; Lateral Extra-articular Tenodesis (LET)
MeSH Terms: conditions — Osteoarthritis; Anterior Cruciate Ligament Injuries; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACL Reconstruction (Active Comparator): Standard ACL reconstruction only.
  Interventions: Procedure: ACL Reconstruction
- ACL + LET (Experimental): Anatomic ACL reconstruction following the same procedure as the active comparator group with an added lateral extra-articular tenodesis (LET).
  Interventions: Procedure: Lateral Extra-Articular Tenodesis (LET); Procedure: ACL Reconstruction

INTERVENTIONS:
Procedure: Lateral Extra-Articular Tenodesis (LET) — Lateral extra-articular tenodesis: A 1cm wide x 8cm long strip of iliotibial band is fashioned, leaving the Gerdys tubercle attachment intact. The graft is tunneled under the fibular collateral ligament (FCL) and attached to the femur with a Richards' staple (Smith & Nephew), just distal to the intermuscular septum, proximal to the femoral insertion of the FCL. Fixation is performed with the knee at 70 degrees flexion, neutral rotation. Minimal tension is applied to the graft. The free end is then looped back onto itself and sutured using the No. 1 vicryl.
  Arms: ACL + LET
Procedure: ACL Reconstruction — Anatomic ACL reconstruction using a four-strand autologous hamstring graft. If the diameter of the graft is found to be less than 7.5mm, semitendinosus will be tripled (5 strand graft) providing a greater graft diameter. Femoral tunnels will be drilled using an anteromedial portal technique, with femoral fixation provided by an Endobutton or equivalent. Tibial fixation will be provided by interference screw.

SUMMARY:
From 2014-2017, across 7 Canadian and 2 European sites, we randomized 618 patients at high-risk of re-injury, to anterior cruciate ligament reconstruction (ACLR) with or without a lateral extraarticular tenodesis (LET) and demonstrated that the addition of the LET reduced the risk of instability (RRR=0.38; 95% Confidence Interval (CI), 0.21-0.52; P=0.0001) and graft re-rupture (RRR, 0.67; 95% CI, 0.36-0.83; P=0.001). As a result, practice has changed; there has been a large increase in the proportion of orthopaedic surgeons recommending the addition of an LET at the time of ACLR and an increase in the number of patients requesting an LET from their surgeon. There is some weak evidence suggesting that in the longer term, the LET may increase the risk of developing osteoarthritis (OA) in that knee. Knee OA affects over 4.4 million Canadians and the number of younger adults being diagnosed with knee OA is growing and is a primary reason for seeking healthcare in Canada. The impact of OA in Canada is enormous and projected to cost Canada $17.5 billion annually in lost productivity alone by 2031. This study will use imaging and patient-reported Knee Outcomes Osteoarthritis Score (KOOS) to evaluate the incidence of OA at 10-years post ACL reconstruction with and without LET. We will also collect information about overall knee health, patient-reported outcomes, costs associated with knee injury, rehabilitation and disability, clinical failure, functional ability, and sport participation. It is crucial that we understand the risks of developing knee OA associated with the addition of an LET to an ACLR so that surgeons and patients can make informed decisions, not just for their immediate post injury treatment of the failed ligament, but for the potential long-term consequences of that decision.

ELIGIBILITY:
Inclusion criteria:

* ACL deficient knee
* skeletally mature to 25 years of age
* 2 or more of:

  * competitive pivoting sport
  * grade 2 pivot shift or greater
  * generalized ligament laxity - Beighton score of 4 or greater

Exclusion criteria:

* previous ACL reconstruction on either knee
* multi-ligament injury (two or more ligaments requiring surgical attention)
* symptomatic articular cartilage defect requiring treatment other than debridement
* greater than 3 degrees of asymmetric varus
* unable to complete outcome questionnaires

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 510 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Lateral compartment knee OA | 10 Years
  As was conducted at baseline and two years postoperative in the Stability 1 study, patients will undergo a standing semi-flexed posterior to anterior (PA) radiograph of both knees.
Region-specific quality of life using the Knee Osteoarthritis and outcomes Score (KOOS) | 10 Years
  The KOOS is a 42-item knee-specific questionnaire with five separately reported domains, including pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sports/recreation (5 items) and knee-related quality of life (4 items). Domain scores represent the average of all items in the domain standardized to a score from 0 to 100 (worst to best). This instrument has face validity and has demonstrated construct validity, excellent test-retest reliability for each domain (range, 0.75 to 0.93) and has been shown to be responsive to change in patients undergoing ACLR.

SECONDARY OUTCOMES:
Disease-specific quality of life using the ACL Quality of Life Questionnaire (ACL-QOL) | 10 Years
  The ACL-QOL has five domains that query physical symptoms, occupational concerns, recreational activities, lifestyle, and social and emotional aspects. Each item has one 100 mm visual analogue scale response option, with labeled anchors at 0 mm (e.g., extremely difficult) and 100 mm (e.g., not difficult at all). Scores are calculated by converting the average of each of the five domain scores to a total average score out of 100% where 100% represents the best possible score.
The Marx Activity Rating Scale (MARS) | 10 Years
  The MARS Activity Rating Scale is a four-item activity rating scale. The patient is asked to rate how often they were able to perform each activity (e.g. running, cutting, decelerating, and pivoting) in their most healthy and active state. The patient is provided with five categories of frequency of each functional activity, ranging from less than one time in a month to four or more times in a week. One point is allocated for each category of frequency and a maximum score of 16 points can be awarded. The MARS has demonstrated excellent test-retest reliability and construct validity in patients with disorders of the knee.
Subjective symptoms, function and activity (IKDC) | 10 Years
  The International Knee Documentation Committee Subjective Knee Form (IKDC) is a knee-specific functional outcome that consists of 18-items about symptoms (7 items), sports activities (10 items) and function (1 item). Likert scales, a dichotomized item and 11 point rating scales make up the response options, and total score ranges from 0 (total limitation) and 100 (no limitations). The IKDC has shown test-retest reliability and good construct validity in patients with issues at the knee.
MRI | 10 Years
  MRI will be performed only on patients recruited from the lead site at the Fowler Kennedy Sport Medicine Clinic (n=196). Similar to the imaging protocol used at the two-year visit, patients will undergo bilateral 3 Tesla MRI on a Siemens Magneton Trio magnet, and a 15-channel Siemens PRISMA knee coil at the 10-year visit. Longer T1rho and T2 relaxation times have shown to be associated with worsening cartilage quality. These changes can also be seen prior to the development of radiographic changes of OA, therefore, MRI can be used as a method for early detection of degenerative changes. The high incidence of arthritic changes observable at the 10 year time point using MRI (compared to plain radiographs), justifies the use of MRI in the subgroup of patients at the lead site.
Patient Reported Quality of Life (ACL QOL) | 10 Years
  The ACL-QOL has five domains that query physical symptoms, occupational concerns, recreational activities, lifestyle, and social and emotional aspects.
  Each item has one 100 mm visual analogue scale response option, with labeled anchors at 0 mm (e.g., extremely difficult) and 100 mm (e.g., not difficult at all). Scores are calculated by converting the average of each of the five domain scores to a total average score out of 100% where 100% represents the best possible score. The ACL-QOL has demonstrated validity in patients with ACL injury and responsiveness to change in patients following ACLR.
4-Item Pain Intensity Measure (P4) | 10 Years
  Four-item questionnaire that asks patients to report the amount of pain they experience throughout the day (morning, afternoon, evening) and with activity. Each item response is a visual analog scale ranging from 0 (no pain) to 10 (as bad as it can be). The total score is a sum of the four responses to a maximum score of 40. The P4 has demonstrated good test-retest reliability and the ability to detect changes in pain intensity in patients with muscle and joint injuries. Because men and women may experience and report pain differently, we have included the Gender Role Expectation of Pain questionnaire to examine its association with pain and quality of life reporting in this study.
Clinical Failure | 10 Years
  As previously described, clinical failure is defined as a composite of symptomatic instability requiring revision ACL surgery, or symptomatic instability with positive pivot shift, or asymmetrical pivot shift greater than the contralateral side.
Objective Functional Measures | 10 Years
  Range of motion (ROM) measurement will include passive knee extension and active-assisted knee flexion. For passive knee extension, the patient is seated with legs extended on a table, heel propped so that the calf and upper thigh clear the treatment table. We will instruct the patient to relax both quadriceps and hamstrings to assure passive measurement. For active assisted knee flexion, the patient is seated with both legs extended on a table. We will instruct them to perform active-assisted knee flexion by placing one hand under their thigh to initiate flexion and then clasp both hands just below the tibial tuberosity. We will measure flexion and extension in degrees using a goniometer. For both measurements, we will centre the fulcrum of the goniometer over the lateral epicondyle of the femur. We will then align the stationary arm of the goniometer with the greater trochanter of the femur and the moving arm with the lateral malleolus at the ankle.
Adverse Events | 10 Years
  We will record adverse events including painful hardware, graft rupture, and reasons for re-operation (e.g., painful knee joint, meniscal injuries, ACLR revision, contralateral ACLR, etc.). Given the significance of these types of events, we expect excellent recall.

CONTACTS AND LOCATIONS:
Locations (8):
- Canada (7):
  - Banff Sport Medicine Clinic, Banff, Alberta
  - University of Calgary, Calgary, Alberta
  - Fraser Health Authority, New Westminster, British Columbia
  - Pan Am Clinic, Winnipeg, Manitoba
  - McMaster University, Hamilton, Ontario
  - Queens University, Kingston, Ontario
  - Fowler Kennedy Sport Medicine Clinic, London, Ontario
- University Hospitals Coventry and Warwickshire NHS Trust, Coventry, United Kingdom